CLINICAL TRIAL: NCT00712244
Title: DisCoVisc Versus Competitor
Brief Title: DisCoVisc Versus DuoVisc, Healon5 and AmVisc Plus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin, Alcon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M07-014
Record Dates: First submitted 2008-07-07; First posted 2008-07-09 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Cataract
Keywords: Discovisc; Ophthalmic Viscosurgical Device
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- DisCoVisc (Active Comparator): Use of DisCoVisc Ophthalmic Viscosurgical Device during cataract surgery.
  Interventions: Device: DisCoVisc
- DuoVisc (Active Comparator): Use of DuoVisc Viscoelastic System (Viscoat, Provisc) during cataract surgery.
  Interventions: Device: DuoVisc
- Healon5 (Active Comparator): Use of Healon5 ophthalmic viscosurgical device (OVD) during cataract surgery.
  Interventions: Device: Healon5
- Amvisc Plus (Active Comparator): Use of Amvisc Plus ophthalmic viscosurgical device during cataract surgery.
  Interventions: Device: Amvisc Plus

INTERVENTIONS:
Device: DisCoVisc — Use of DisCoVisc Ophthalmic Viscosurgical Device (4% sodium chondroitin sulfate, 1.65% sodium hyaluronate) during cataract surgery.
  Arms: DisCoVisc
Device: DuoVisc — Use of DuoVisc viscoelastic system consisting of Viscoat (3% sodium hyaluronate, 4% chondroitin sulfate)and Provisc(1% sodium hyaluronate) during cataract surgery.
  Arms: DuoVisc
Device: Healon5 — Use of Healon5 ophthalmic viscosurgical device (2.3% Sodium Hyaluronate) during cataract surgery.
  Arms: Healon5
Device: Amvisc Plus — Use of Amvisc Plus ophthalmic viscosurgical device (1.6% Sodium Hyaluronate) during cataract surgery.
  Arms: Amvisc Plus

SUMMARY:
A comparison of the ability of DisCoVisc to that of other ophthalmic viscosurgical devices (OVDs) (DuoVisc, Healon5 or Amvisc PLUS) regarding endothelial protection and anterior chamber space maintenance during non-eventful cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* operable cataracts in at least one eye

Exclusion Criteria:

* Endothelial Cell Count (ECC) ≤1500cells/mm2
* Intraocular Pressure (IOP) > 21mm Hg
* previous ocular inflammation
* systemic or ocular conditions affecting corneal endothelium

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Study Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were >50 years old & of any race & gender. Subjects had operable cataracts in at least 1 eye, were able to provide informed consent, & were free of systemic diseases affecting ocular health, especially those affecting endothelial cell counts. Eyes were free of ocular disease & had no history of chronic/recurrent inflammatory eye disease.
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study by meeting all inclusion/exclusion criteria were enrolled. Group assignment was based on an Excel randomization scheme.
Groups:
- DISCOVISC: DISCOVISC® Ophthalmic Viscosurgical Device (OVD)
- DUOVISC: DUOVISC® Viscoelastic system
- Healon5: Healon5 Ophthalmic Viscosurgical Device
- Amvisc Plus: Amvisc Plus Ophthalmic Viscosurgical Device
Period: Overall Study
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Started | 29 | 29 | 27 | 27
Completed | 25 | 28 | 25 | 26
Not Completed | 4 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus | Total
Number analyzed (Participants) | 29 | 29 | 27 | 27 | 112
Age Categorical [Number; unit: participants] — Age data not available for 2 DisCoVisc subjects, 2 Duovisc subjects, and 1 AmVisc Plus subject.
  participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 12 | 12 | 9 | 8 | 41
    >=65 years | 16 | 15 | 18 | 18 | 67
Gender [Number; unit: participants] — Gender not available for 2 DisCoVisc subjects, 1 Duovisc subject, and 1 AmVisc Plus subject.
  participants
    Female | 18 | 15 | 16 | 19 | 68
    Male | 10 | 12 | 11 | 7 | 40

OUTCOME MEASURES:

1. Primary Outcome: Corneal Endothelial Cell Loss
Description: Percentage of corneal endothelial cells lost 1 month after surgery as compared to the number of corneal endothelial cells measured before surgery. Corneal endothelial cells are measured by counting the number of cells on an image taken by specular microscope.
Time Frame: 1 month after surgery
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 24 | 26 | 24 | 25
Percent Change | 1.51 (5.99) | 1.18 (11.18) | 4.72 (7.23) | 6.30 (14.31)

2. Secondary Outcome: Percent Gain in Corneal Thickness.
Description: Percent Gain in Corneal Thickness between the assessment performed before surgery to that performed after surgery. This was assessed at both the 1 week and 1 month visit. Corneal thickness is measured in micrometers and is evaluated by Pachymetry. A negative number indicates a decrease in corneal thickness.
Time Frame: 1 week and month after surgery
Population: Participants analyzed for Baseline to 1 week: 29 DisCovisc, 28 DuoVisc, 26 Healon5, 26 Amvisc Plus.
Measure: Mean (Standard Deviation); unit: Percent Gain
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 25 | 28 | 25 | 26
Percent Gain
  Before Surgery to 1 Week after Surgery | 2.89 (16.45) | 7.02 (12.06) | 9.92 (15.29) | 5.06 (12.07)
  Before Surgery to 1 Month after Surgery | -0.55 (11.79) | -1.06 (25.38) | 1.98 (10.57) | -9.11 (22.85)

3. Secondary Outcome: Aqueous Signs - Corneal Edema
Description: Measured as the percentage of patient's eyes subjectively evaluated to have corneal edema at each of the following gradings: 0 - none; 1 - Mild, slight localized or generalized edema; 2 - Moderate, significant localized or generalized edema; 3 - Severe, advanced localized or generalized edema.
Time Frame: 1 day after surgery
Population: This data was collected for all subjects attending the visit one day after surgery.
Measure: Number; unit: Percentage of Participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 26 | 26
Percentage of Participants
  None | 68.97 | 75 | 57.69 | 65.38
  Mild | 57.59 | 21.43 | 34.62 | 34.62
  Moderate | 3.45 | 3.57 | 7.69 | 0
  Severe | 0 | 0 | 0 | 0

4. Secondary Outcome: Aqueous Signs - Aqueous Flare
Description: Measured as the percentage of patient's eyes subjectively evaluated to have Aqueous Flare at each of the following gradings: 0 - None: No visible flare when compared to the normal eye, 1 - Mild: Flare visible against dark papillary background but not visible against iris background, 2 - Moderate: Flare is visible with the slit-lamp beam aimed onto the iris surface as well as teh dark papillary background, 3 - Severe: Very dense flare. May also present as a hazy appearance of anterior segment structures when viewed with low power magnification of the slit-lamp.
Time Frame: 1 Day after Surgery
Population: This data was collected for all subjects attending the visit one day after surgery.
Measure: Number; unit: Percentage of participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 26 | 26
Percentage of participants
  None | 20.69 | 39.29 | 26.92 | 46.15
  Mild | 75.86 | 53.57 | 65.38 | 53.85
  Moderate | 3.45 | 7.14 | 7.69 | 0
  Severe | 0 | 0 | 0 | 0

5. Secondary Outcome: Aqueous Signs - Aqueous Cells
Description: Measured as the percentage of patient's eyes subjectively evaluated to have Aqueous Cells at each of the following gradings: 0 - None, 1 - 1 to 5 cells, 2 - 6 to 15 cells, 3 - 16 - 30 cells, 4 - >30 cells.
Time Frame: 1 day after surgery
Population: This data was collected for all subjects attending the visit one day after surgery.
Measure: Number; unit: Percentage of participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 26 | 26
Percentage of participants
  Grade 0 | 6.9 | 14.29 | 7.69 | 7.69
  Grade 1 | 65.52 | 46.43 | 50 | 65.38
  Grade 2 | 24.14 | 32.14 | 38.46 | 23.08
  Grade 3 | 3.45 | 7.14 | 3.85 | 3.85
  Grade 4 | 0 | 0 | 0 | 0

6. Secondary Outcome: Intraocular Pressure (IOP)
Description: Measure of intraocular pressure of a patient's eye via tonometry one day after surgery. Measured in mmHg. Normal intraocular pressure is between 10 mmHg and 20 mmHg.
Time Frame: 1 day after surgery
Population: This data was collected on all subjects attending the visit one day after surgery with the exception of 3 DisCoVisc subjects, 4 DuoVisc subjects, 2 Healon5 subjects, and 1 AmVisc Plus subject.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 26 | 25 | 25 | 26
mmHg | 21.58 (8.42) | 19.48 (4.6) | 20.72 (6.61) | 18.65 (5.56)

7. Secondary Outcome: Surgeon Survey - Anterior Chamber Dome Maintenance During Anterior Capsulotomy
Description: Surgeon reporting of Anterior Chamber Dome Maintenance of a subject's eye during anterior capsulotomy. Evaluated on a subjective scale and reported as percent by response. The following scale is used, from worst to best: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance.
Time Frame: Time of surgery
Population: This data was collected on all subjects undergoing surgery with the exception of 1 DuoVisc subject.
Measure: Number; unit: Percentage of participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 27 | 27
Percentage of participants
  Flat | 0 | 0 | 0 | 0
  Shallow | 3.45 | 3.57 | 22.22 | 18.52
  Working Space Adequate | 0 | 7.14 | 48.15 | 55.56
  Full Chamber Maintenance | 96.55 | 89.29 | 29.63 | 25.93

8. Secondary Outcome: Surgeon Surgey - Anterior Dome Maintenance During Phacoemulsification
Description: Surgeon reporting of Anterior Chamber Dome Maintenance of a subject's eye during phacoemulsification. Evaluated on a subjective scale and reported as percent by response. The following scale is used, from worst to best: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance.
Time Frame: Time of Surgery
Population: This data was collected on all subjects undergoing surgery with the exception of 1 DuoVisc subject.
Measure: Number; unit: Percentage of participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 27 | 27
Percentage of participants
  Flat | 0 | 0 | 0 | 0
  Shallow | 0 | 0 | 11.11 | 3.7
  Working Space Adequate | 0 | 3.57 | 51.85 | 48.15
  Full Chamber Maintenance | 100 | 96.43 | 37.04 | 48.15

9. Secondary Outcome: Surgeon Surgey - Anterior Dome Maintenance During Intraocular Lens (IOL) Insertion
Description: Surgeon reporting of Anterior Chamber Dome Maintenance of a subject's eye during intraocular lens (IOL) insertion. Evaluated on a subjective scale and reported as percent by response. The following scale is used, from worst to best: Flat, Shallow, Working Space Adequate, Full Chamber Maintenance.
Time Frame: Time of Surgery
Population: This data was collected on all subjects undergoing surgery with the exception of 1 DuoVisc subject.
Measure: Number; unit: Percentage of participants
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Number analyzed (Participants) | 29 | 28 | 27 | 27
Percentage of participants
  Flat | 0 | 0 | 0 | 0
  Shallow | 0 | 0 | 40.74 | 7.41
  Working Space Adequate | 0 | 7.14 | 25.93 | 44.44
  Full Chamber Maintenance | 100 | 92.86 | 33.33 | 48.15

ADVERSE EVENTS:
Description: There were no adverse events reported for this study.
Arm/Group | DISCOVISC | DUOVISC | Healon5 | Amvisc Plus
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/27 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.